CLINICAL TRIAL: NCT05853848
Title: Randomized Comparison of Mail- and Phone-based Interventions Promoting Mammogram Screening
Brief Title: Mammogram Mail- and Phone-based Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-0369
Record Dates: First submitted 2023-04-28; First posted 2023-05-11 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Economics, Behavioral; Mammography; Risk Reduction Behavior; Communication
MeSH Terms: conditions — Breast Neoplasms; Behavior; Risk Reduction Behavior; Communication | interventions — College Fraternities and Sororities

STUDY DESIGN:
Intervention Model Description: Each intervention will be rolled out to only a subset of the total population each month, such that all patients will receive one of the interventions over the course of 7 months. Active arms will be compared contemporaneously against a passive control group consisting of active arm participants for whom the intervention has not yet begun, as well as a random subset of participants who are excluded before the future intervention begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard postcard (Active Comparator): Patients in this arm will receive a postcard with words and an image, typical of outreach in prior years, encouraging them to schedule their annual mammograms.
  Interventions: Behavioral: Postcard
- Formal letter (Experimental): Patients in this arm will receive a letter from the Geisinger Health Plan (on Geisinger letterhead) noting that they're overdue for a mammogram and encouraging them to schedule.
  Interventions: Behavioral: Letter
- Auto-dialer (Experimental): Patients in this arm will receive a call from an auto-dialer with a message noting that they're overdue for a mammogram and encouraging them to schedule.
  Interventions: Behavioral: Auto-dialer
- Live call (Experimental): Patients in this arm will receive a call from a Geisinger Health Plan representative noting that they're overdue for a mammogram and encouraging them to schedule (and helping them schedule if they are interested).
  Interventions: Behavioral: Live call

INTERVENTIONS:
Behavioral: Postcard — Postcard with phone number to call for help scheduling a mammogram.
  Arms: Standard postcard
Behavioral: Letter — Letter with phone number to call for help scheduling a mammogram.
  Arms: Formal letter
Behavioral: Auto-dialer — Auto-dialer with option to press button for help scheduling a mammogram.
  Arms: Auto-dialer
Behavioral: Live call — Live call offering help scheduling a mammogram.
  Arms: Live call

SUMMARY:
The project aims to evaluate four different versions and modalities of interventions encouraging mammogram screening among all eligible women due or overdue for screening. The evaluation will compare among the following forms of outreach to help determine whether (a) live calls are more effective at increasing mammogram screening than other forms of outreach and (b) each form of outreach is more effective than no outreach: (1) a postcard, (2) a letter, (3) an auto-dialer phone message, and (4) a live call from a care gaps team. The interventions will be rolled out over many months, allowing for comparisons of effectiveness against those who have not yet been contacted.

ELIGIBILITY:
Inclusion Criteria:

* Female Geisinger Health Plan members between ages 52 and 74 as of December 31, 2023
* Overdue for annual mammogram
* Continuously enrolled with the Geisinger Health Plan as of October 1, 2021
* Can be contacted via both phone and mail

Exclusion Criteria:

* Geisinger Health Plan members on a do-not-contact list
* Had a mammogram as of October 1, 2021
* In hospice, using hospice services, or receiving palliative care as of January 1, 2023
* Medicare members 66 years of age or above at time of outreach, who are institutionalized or have both frailty and advanced illness
* Had a bilateral mastectomy at any time

Ages: 51 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14386 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Mammogram completed | In the 180 days following the patient's intervention send date
  Record of completed mammogram (yes/no), for comparing postcards, letters, and auto-dialer messages with live calls
Mammogram completed | In the 120 days following the patient's intervention send date
  Record of completed mammogram (yes/no), for comparing postcards, letters, auto-dialer messages, and live calls with controls

OTHER OUTCOMES:
Mammogram completed | In the 180 days following the patient's intervention send date
  Record of completed mammogram (yes/no), for comparing across postcards, letters, and auto-dialer messages
Breast malignancy risk detected | In the 210 days following the patient's intervention send date
  Record of high malignancy risk (yes/no), for comparing across different modalities of outreach
Mammogram appointment scheduled | In the 30 days following the patient's intervention send date
  Appointment scheduled for mammogram, among patients visiting Geisinger clinics (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: By the paper's online publication date. Data will remain available for as long as the Open Science Framework hosts it.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT05853848/Prot_SAP_000.pdf